CLINICAL TRIAL: NCT04199767
Title: SNIFF Multi-Device Study 2 - Study of Nasal Insulin to Fight Forgetfulness
Brief Title: SNIFF Multi-Device Study 2
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Paused for preliminary data analysis.
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00062612
Record Dates: First submitted 2019-12-12; First posted 2019-12-16 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2024-09

CONDITIONS: Mild Cognitive Impairment; Cognitive Impairment
Keywords: Intranasal Delivery of Insulin; Cognitive Testing; Nasal Insulin
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Commerce

STUDY DESIGN:
Intervention Model Description: At study entry, participants will be randomized to receive either 20 or 40 International Units of insulin first and the opposite substance on a second visit.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Neither participants or site personnel will know which dose of insulin is being administered. Exceptions will be the study nurse who is directly involved in preparing the insulin.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 20 IU Insulin first, then 40 IU Insulin (Experimental): Participants will be randomly assigned to receive regular insulin (U100, 20 IU) administered with an intranasal nebulizer-like device. Participants in this arm will then receive regular insulin (U100, 40 IU) at visit 3 during second intervention period.
  Interventions: Drug: 20 IU Humulin® R U-100 (NDC: 0002-8215, Eli Lilly & Company)
- 40 IU Insulin first, then 20 IU Insulin (Experimental): Participants will be randomly assigned to receive regular insulin (U100, 40 IU) administered with an intranasal nebulizer-like device. Participants in this arm will then receive regular insulin (U100, 20 IU) at visit 3 during second intervention period.
  Interventions: Drug: 40 IU Humulin® R U-100 (NDC: 0002-8215, Eli Lilly & Company)

INTERVENTIONS:
Drug: 20 IU Humulin® R U-100 (NDC: 0002-8215, Eli Lilly & Company) — Participants will be assigned to receive regular insulin either 20 or 40 IU administered through an intranasal nebulizer-like device.
  Other Names: Humulin® R U-100
  Arms: 20 IU Insulin first, then 40 IU Insulin
Drug: 40 IU Humulin® R U-100 (NDC: 0002-8215, Eli Lilly & Company) — Participants will be assigned to receive regular insulin either 40 or 20 IU administered through an intranasal nebulizer-like device.
  Other Names: Humulin® R U-100
  Arms: 40 IU Insulin first, then 20 IU Insulin

SUMMARY:
The SNIFF Device study will involve using one of three devices to administer insulin through each participant's nose or intra-nasally, accompanied by a lumbar puncture. This goal of this study is to measure how much insulin the device delivers to the cerebrospinal fluid (CSF). In addition, this study will look at the effects of insulin administered intra-nasally on memory, and on blood levels of insulin.

DETAILED DESCRIPTION:
The aim of this study is to determine the ability of an intranasal delivery device to increase levels of insulin in cerebrospinal fluid (CSF).

A growing body of evidence suggests that insulin plays a role in normal memory processes and that insulin abnormalities may contribute to cognitive and brain changes associated with Alzheimer's disease (AD). Interestingly, insulin administered to the nasal cavity is transported within a few minutes into the brain, but does not affect blood sugar or insulin levels.

The study will consist of a single site, randomized, double-blind trial comparing the acute effects of INI 20 International Units or 40 International Units delivered with one of three nebulizer-like devices on CSF insulin levels, AD biomarkers and memory. At study entry, participants will be randomized to receive either 20 or 40 IU insulin first, and the opposite dose on a second visit. Participants who are cognitively normal or who have aMCI (n=30) will be enrolled. The primary outcome measure will be to establish which device and which dose provides the greatest increase in CSF insulin which will provide important evidence to be used in the design of future trials.

ELIGIBILITY:
Inclusion Criteria:

* Fluent in English
* Cognitively normal or diagnosis of aMCI
* Stable medical condition for 3 months prior to screening visit
* Stable medications for 4 weeks prior to the screening and study visits
* Clinical laboratory values must be within normal limits or, if abnormal, must be judged to be clinically insignificant by the study physician

Exclusion Criteria:

* A diagnosis of dementia
* History of a clinically significant stroke
* Current evidence or history in past two years of epilepsy, head injury with loss of consciousness, any major psychiatric disorder including psychosis, major depression, bipolar disorder
* Diabetes (type I or type II) insulin dependent and non-insulin dependent diabetes mellitus
* Current or past regular use of insulin or any other anti-diabetic medication within 2 months of screening visit.
* History of seizure within past five years
* Pregnancy or possible pregnancy.
* Use of anticoagulants warfarin (Coumadin) and dabigatran (Pradaxa)
* Residence in a skilled nursing facility at screening
* Use of an investigational agent within two months of screening visit
* Regular use of alcohol, narcotics, anticonvulsants, anti-parkinsonian medications, or any other exclusionary medications

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-07-16 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
CSF insulin levels | 30 minutes after intervention administration
  To compare changes in CSF insulin levels after receiving a 20 or 40 International Unit dose of insulin delivered with one of three devices, compared to baseline levels.

SECONDARY OUTCOMES:
Auditory-Verbal Learning Test (AVLT) | 5 minutes before lumbar puncture, and immediately following lumbar puncture.
  To examine differences in memory performance measured with a list learning test (Auditory Verbal Learning Test) after administration of 20 or 40 IU insulin.

OTHER OUTCOMES:
CSF Levels of AB42 | 30 minutes after intervention administration
  Levels of the 42 amino acid isoform of the beta amyloid peptide

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Craft, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Albert MS, DeKosky ST, Dickson D, Dubois B, Feldman HH, Fox NC, Gamst A, Holtzman DM, Jagust WJ, Petersen RC, Snyder PJ, Carrillo MC, Thies B, Phelps CH. The diagnosis of mild cognitive impairment due to Alzheimer's disease: recommendations from the National Institute on Aging-Alzheimer's Association workgroups on diagnostic guidelines for Alzheimer's disease. Alzheimers Dement. 2011 May;7(3):270-9. doi: 10.1016/j.jalz.2011.03.008. Epub 2011 Apr 21. PMID 21514249
- [Background] Baker H, Spencer RF. Transneuronal transport of peroxidase-conjugated wheat germ agglutinin (WGA-HRP) from the olfactory epithelium to the brain of the adult rat. Exp Brain Res. 1986;63(3):461-73. doi: 10.1007/BF00237470. PMID 3758265
- [Background] Baker LD, Cross DJ, Minoshima S, Belongia D, Watson GS, Craft S. Insulin resistance and Alzheimer-like reductions in regional cerebral glucose metabolism for cognitively normal adults with prediabetes or early type 2 diabetes. Arch Neurol. 2011 Jan;68(1):51-7. doi: 10.1001/archneurol.2010.225. Epub 2010 Sep 13. PMID 20837822
- [Background] Balin BJ, Broadwell RD, Salcman M, el-Kalliny M. Avenues for entry of peripherally administered protein to the central nervous system in mouse, rat, and squirrel monkey. J Comp Neurol. 1986 Sep 8;251(2):260-80. doi: 10.1002/cne.902510209. PMID 3782501
- [Background] Benedict C, Hallschmid M, Hatke A, Schultes B, Fehm HL, Born J, Kern W. Intranasal insulin improves memory in humans. Psychoneuroendocrinology. 2004 Nov;29(10):1326-34. doi: 10.1016/j.psyneuen.2004.04.003. PMID 15288712
- [Background] Benedict C, Kern W, Schultes B, Born J, Hallschmid M. Differential sensitivity of men and women to anorexigenic and memory-improving effects of intranasal insulin. J Clin Endocrinol Metab. 2008 Apr;93(4):1339-44. doi: 10.1210/jc.2007-2606. Epub 2008 Jan 29. PMID 18230654
- [Background] Born J, Lange T, Kern W, McGregor GP, Bickel U, Fehm HL. Sniffing neuropeptides: a transnasal approach to the human brain. Nat Neurosci. 2002 Jun;5(6):514-6. doi: 10.1038/nn849. No abstract available. PMID 11992114
- [Background] Bodian, D. and H. A. Howe (1941).
- [Background] Broadwell RD, Balin BJ. Endocytic and exocytic pathways of the neuronal secretory process and trans-synaptic transfer of wheat germ agglutinin-horseradish peroxidase in vivo. J Comp Neurol. 1985 Dec 22;242(4):632-50. doi: 10.1002/cne.902420410. PMID 2418083
- [Background] Cavanna AE, Trimble MR. The precuneus: a review of its functional anatomy and behavioural correlates. Brain. 2006 Mar;129(Pt 3):564-83. doi: 10.1093/brain/awl004. Epub 2006 Jan 6. PMID 16399806
- [Background] Chiu SL, Chen CM, Cline HT. Insulin receptor signaling regulates synapse number, dendritic plasticity, and circuit function in vivo. Neuron. 2008 Jun 12;58(5):708-19. doi: 10.1016/j.neuron.2008.04.014. PMID 18549783
- [Background] Craft S, Baker LD, Montine TJ, Minoshima S, Watson GS, Claxton A, Arbuckle M, Callaghan M, Tsai E, Plymate SR, Green PS, Leverenz J, Cross D, Gerton B. Intranasal insulin therapy for Alzheimer disease and amnestic mild cognitive impairment: a pilot clinical trial. Arch Neurol. 2012 Jan;69(1):29-38. doi: 10.1001/archneurol.2011.233. Epub 2011 Sep 12. PMID 21911655
- [Background] Craft S, Peskind E, Schwartz MW, Schellenberg GD, Raskind M, Porte D Jr. Cerebrospinal fluid and plasma insulin levels in Alzheimer's disease: relationship to severity of dementia and apolipoprotein E genotype. Neurology. 1998 Jan;50(1):164-8. doi: 10.1212/wnl.50.1.164. PMID 9443474
- [Background] Craft S, Watson GS. Insulin and neurodegenerative disease: shared and specific mechanisms. Lancet Neurol. 2004 Mar;3(3):169-78. doi: 10.1016/S1474-4422(04)00681-7. PMID 14980532
- [Background] De Felice FG, Vieira MN, Bomfim TR, Decker H, Velasco PT, Lambert MP, Viola KL, Zhao WQ, Ferreira ST, Klein WL. Protection of synapses against Alzheimer's-linked toxins: insulin signaling prevents the pathogenic binding of Abeta oligomers. Proc Natl Acad Sci U S A. 2009 Feb 10;106(6):1971-6. doi: 10.1073/pnas.0809158106. Epub 2009 Feb 2. PMID 19188609
- [Background] Faber, H. K. (1938).
- [Background] Fairbrother, R. W. and E. W. Hurst (1930).
- [Background] Fishel MA, Watson GS, Montine TJ, Wang Q, Green PS, Kulstad JJ, Cook DG, Peskind ER, Baker LD, Goldgaber D, Nie W, Asthana S, Plymate SR, Schwartz MW, Craft S. Hyperinsulinemia provokes synchronous increases in central inflammation and beta-amyloid in normal adults. Arch Neurol. 2005 Oct;62(10):1539-44. doi: 10.1001/archneur.62.10.noc50112. PMID 16216936
- [Background] Francis GJ, Martinez JA, Liu WQ, Xu K, Ayer A, Fine J, Tuor UI, Glazner G, Hanson LR, Frey WH 2nd, Toth C. Intranasal insulin prevents cognitive decline, cerebral atrophy and white matter changes in murine type I diabetic encephalopathy. Brain. 2008 Dec;131(Pt 12):3311-34. doi: 10.1093/brain/awn288. Epub 2008 Nov 16. PMID 19015157 (Retraction: PMID 24860127 Brain. 2014 Jun;137(Pt 6):e283)
- [Background] Frolich L, Blum-Degen D, Bernstein HG, Engelsberger S, Humrich J, Laufer S, Muschner D, Thalheimer A, Turk A, Hoyer S, Zochling R, Boissl KW, Jellinger K, Riederer P. Brain insulin and insulin receptors in aging and sporadic Alzheimer's disease. J Neural Transm (Vienna). 1998;105(4-5):423-38. doi: 10.1007/s007020050068. PMID 9720972
- [Background] Galasko D, Bennett D, Sano M, Ernesto C, Thomas R, Grundman M, Ferris S. An inventory to assess activities of daily living for clinical trials in Alzheimer's disease. The Alzheimer's Disease Cooperative Study. Alzheimer Dis Assoc Disord. 1997;11 Suppl 2:S33-9. PMID 9236950
- [Background] Gasparini L, Gouras GK, Wang R, Gross RS, Beal MF, Greengard P, Xu H. Stimulation of beta-amyloid precursor protein trafficking by insulin reduces intraneuronal beta-amyloid and requires mitogen-activated protein kinase signaling. J Neurosci. 2001 Apr 15;21(8):2561-70. doi: 10.1523/JNEUROSCI.21-08-02561.2001. PMID 11306609
- [Background] Gil-Bea FJ, Solas M, Solomon A, Mugueta C, Winblad B, Kivipelto M, Ramirez MJ, Cedazo-Minguez A. Insulin levels are decreased in the cerebrospinal fluid of women with prodomal Alzheimer's disease. J Alzheimers Dis. 2010;22(2):405-13. doi: 10.3233/JAD-2010-100795. PMID 20847404
- [Background] Hallschmid M, Benedict C, Schultes B, Born J, Kern W. Obese men respond to cognitive but not to catabolic brain insulin signaling. Int J Obes (Lond). 2008 Feb;32(2):275-82. doi: 10.1038/sj.ijo.0803722. Epub 2007 Sep 11. PMID 17848936
- [Background] Hong M, Lee VM. Insulin and insulin-like growth factor-1 regulate tau phosphorylation in cultured human neurons. J Biol Chem. 1997 Aug 1;272(31):19547-53. doi: 10.1074/jbc.272.31.19547. PMID 9235959
- [Background] Hughes CP, Berg L, Danziger WL, Coben LA, Martin RL. A new clinical scale for the staging of dementia. Br J Psychiatry. 1982 Jun;140:566-72. doi: 10.1192/bjp.140.6.566. PMID 7104545
- [Background] Illum L. Nasal drug delivery: new developments and strategies. Drug Discov Today. 2002 Dec 1;7(23):1184-9. doi: 10.1016/s1359-6446(02)02529-1. PMID 12547019
- [Background] Kern W, Born J, Schreiber H, Fehm HL. Central nervous system effects of intranasally administered insulin during euglycemia in men. Diabetes. 1999 Mar;48(3):557-63. doi: 10.2337/diabetes.48.3.557. PMID 10078556
- [Background] Kristensson K, Olsson Y. Uptake of exogenous proteins in mouse olfactory cells. Acta Neuropathol. 1971;19(2):145-54. doi: 10.1007/BF00688493. No abstract available. PMID 5126829
- [Background] Kupila A, Sipila J, Keskinen P, Simell T, Knip M, Pulkki K, Simell O. Intranasally administered insulin intended for prevention of type 1 diabetes--a safety study in healthy adults. Diabetes Metab Res Rev. 2003 Sep-Oct;19(5):415-20. doi: 10.1002/dmrr.397. PMID 12951650
- [Background] Lee CC, Kuo YM, Huang CC, Hsu KS. Insulin rescues amyloid beta-induced impairment of hippocampal long-term potentiation. Neurobiol Aging. 2009 Mar;30(3):377-87. doi: 10.1016/j.neurobiolaging.2007.06.014. Epub 2007 Aug 10. PMID 17692997
- [Background] Minoshima S, Frey KA, Foster NL, Kuhl DE. Preserved pontine glucose metabolism in Alzheimer disease: a reference region for functional brain image (PET) analysis. J Comput Assist Tomogr. 1995 Jul-Aug;19(4):541-7. doi: 10.1097/00004728-199507000-00006. PMID 7622680
- [Background] Minoshima S, Koeppe RA, Frey KA, Kuhl DE. Anatomic standardization: linear scaling and nonlinear warping of functional brain images. J Nucl Med. 1994 Sep;35(9):1528-37. PMID 8071705
- [Background] Morris JC, Ernesto C, Schafer K, Coats M, Leon S, Sano M, Thal LJ, Woodbury P. Clinical dementia rating training and reliability in multicenter studies: the Alzheimer's Disease Cooperative Study experience. Neurology. 1997 Jun;48(6):1508-10. doi: 10.1212/wnl.48.6.1508. PMID 9191756
- [Background] Petersen RC, Doody R, Kurz A, Mohs RC, Morris JC, Rabins PV, Ritchie K, Rossor M, Thal L, Winblad B. Current concepts in mild cognitive impairment. Arch Neurol. 2001 Dec;58(12):1985-92. doi: 10.1001/archneur.58.12.1985. PMID 11735772
- [Background] Pontiroli AE, Alberetto M, Secchi A, Dossi G, Bosi I, Pozza G. Insulin given intranasally induces hypoglycaemia in normal and diabetic subjects. Br Med J (Clin Res Ed). 1982 Jan 30;284(6312):303-6. doi: 10.1136/bmj.284.6312.303. PMID 6800439
- [Background] Reger MA, Watson GS, Frey WH 2nd, Baker LD, Cholerton B, Keeling ML, Belongia DA, Fishel MA, Plymate SR, Schellenberg GD, Cherrier MM, Craft S. Effects of intranasal insulin on cognition in memory-impaired older adults: modulation by APOE genotype. Neurobiol Aging. 2006 Mar;27(3):451-8. doi: 10.1016/j.neurobiolaging.2005.03.016. Epub 2005 Jun 16. PMID 15964100
- [Background] Reger MA, Watson GS, Green PS, Baker LD, Cholerton B, Fishel MA, Plymate SR, Cherrier MM, Schellenberg GD, Frey WH 2nd, Craft S. Intranasal insulin administration dose-dependently modulates verbal memory and plasma amyloid-beta in memory-impaired older adults. J Alzheimers Dis. 2008 Apr;13(3):323-31. doi: 10.3233/jad-2008-13309. PMID 18430999
- [Background] Reger MA, Watson GS, Green PS, Wilkinson CW, Baker LD, Cholerton B, Fishel MA, Plymate SR, Breitner JC, DeGroodt W, Mehta P, Craft S. Intranasal insulin improves cognition and modulates beta-amyloid in early AD. Neurology. 2008 Feb 5;70(6):440-8. doi: 10.1212/01.WNL.0000265401.62434.36. Epub 2007 Oct 17. PMID 17942819
- [Background] Rivera EJ, Goldin A, Fulmer N, Tavares R, Wands JR, de la Monte SM. Insulin and insulin-like growth factor expression and function deteriorate with progression of Alzheimer's disease: link to brain reductions in acetylcholine. J Alzheimers Dis. 2005 Dec;8(3):247-68. doi: 10.3233/jad-2005-8304. PMID 16340083
- [Background] Rubin, D. B. (1987). Multiple Imputation for Nonresponse in Surveys. Hoboken, New Jersey, John Wiley & Sons, Inc
- [Background] Sakane T, Akizuki M, Taki Y, Yamashita S, Sezaki H, Nadai T. Direct drug transport from the rat nasal cavity to the cerebrospinal fluid: the relation to the molecular weight of drugs. J Pharm Pharmacol. 1995 May;47(5):379-81. doi: 10.1111/j.2042-7158.1995.tb05814.x. PMID 7494186
- [Background] Sano M, Raman R, Emond J, Thomas RG, Petersen R, Schneider LS, Aisen PS. Adding delayed recall to the Alzheimer Disease Assessment Scale is useful in studies of mild cognitive impairment but not Alzheimer disease. Alzheimer Dis Assoc Disord. 2011 Apr-Jun;25(2):122-7. doi: 10.1097/WAD.0b013e3181f883b7. PMID 20921876
- [Background] Selkoe DJ. Soluble oligomers of the amyloid beta-protein impair synaptic plasticity and behavior. Behav Brain Res. 2008 Sep 1;192(1):106-13. doi: 10.1016/j.bbr.2008.02.016. Epub 2008 Feb 17. PMID 18359102
- [Background] Shipley MT. Transport of molecules from nose to brain: transneuronal anterograde and retrograde labeling in the rat olfactory system by wheat germ agglutinin-horseradish peroxidase applied to the nasal epithelium. Brain Res Bull. 1985 Aug;15(2):129-42. doi: 10.1016/0361-9230(85)90129-7. PMID 3840049
- [Background] Stockhorst U, de Fries D, Steingrueber HJ, Scherbaum WA. Insulin and the CNS: effects on food intake, memory, and endocrine parameters and the role of intranasal insulin administration in humans. Physiol Behav. 2004 Oct 30;83(1):47-54. doi: 10.1016/j.physbeh.2004.07.022. PMID 15501490
- [Background] Thorne RG, Emory CR, Ala TA, Frey WH 2nd. Quantitative analysis of the olfactory pathway for drug delivery to the brain. Brain Res. 1995 Sep 18;692(1-2):278-82. doi: 10.1016/0006-8993(95)00637-6. PMID 8548316
- [Background] Thorne RG, Pronk GJ, Padmanabhan V, Frey WH 2nd. Delivery of insulin-like growth factor-I to the rat brain and spinal cord along olfactory and trigeminal pathways following intranasal administration. Neuroscience. 2004;127(2):481-96. doi: 10.1016/j.neuroscience.2004.05.029. PMID 15262337
- [Background] Townsend M, Mehta T, Selkoe DJ. Soluble Abeta inhibits specific signal transduction cascades common to the insulin receptor pathway. J Biol Chem. 2007 Nov 16;282(46):33305-33312. doi: 10.1074/jbc.M610390200. Epub 2007 Sep 13. PMID 17855343
- [Background] Weiss P, Holland Y. Neuronal dynamics and axonal flow, ii. The olfactory nerve as model test object. Proc Natl Acad Sci U S A. 1967 Feb;57(2):258-64. doi: 10.1073/pnas.57.2.258. No abstract available. PMID 16591462
- [Background] Worsley KJ, Evans AC, Marrett S, Neelin P. A three-dimensional statistical analysis for CBF activation studies in human brain. J Cereb Blood Flow Metab. 1992 Nov;12(6):900-18. doi: 10.1038/jcbfm.1992.127. PMID 1400644
- [Background] Zhao L, Teter B, Morihara T, Lim GP, Ambegaokar SS, Ubeda OJ, Frautschy SA, Cole GM. Insulin-degrading enzyme as a downstream target of insulin receptor signaling cascade: implications for Alzheimer's disease intervention. J Neurosci. 2004 Dec 8;24(49):11120-6. doi: 10.1523/JNEUROSCI.2860-04.2004. PMID 15590928
- [Background] Zhao WQ, Townsend M. Insulin resistance and amyloidogenesis as common molecular foundation for type 2 diabetes and Alzheimer's disease. Biochim Biophys Acta. 2009 May;1792(5):482-96. doi: 10.1016/j.bbadis.2008.10.014. Epub 2008 Nov 5. PMID 19026743